CLINICAL TRIAL: NCT07374224
Title: A Phase I, Open-label, Two-part, Fixed-sequence Drug Interaction Study to Evaluate the Effects of Concomitant Use of the CYP3A4 Inhibitor Itraconazole or the CYP3A4 Inducer Rifampin on the Pharmacokinetics of Rocbrutinib in Healthy Subjects
Brief Title: A Study Evaluating the Effects of Itraconazole or Rifampin on the Pharmacokinetic Characteristics of Rocbrutinib Tablet
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN107
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Clinical Pharmacology
Keywords: drug interaction; Rocbrutinib; LP-168; CYP3A4
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhibitor Group (Experimental): The Inhibitor Group was designed to investigate the drug-drug interaction between Rocbrutinib and itraconazole (a potent CYP3A inhibitor and P-gp inhibitor). Itraconazole is a recommended potent index CYP3A inhibitor for clinical studies in the ICH-M12 Guideline on Drug Interactions. In accordance with the recommendations in an industry white paper (CPT Pharmacometrics Syst Pharmacol. 2019 Aug 7;8(9):685-695), an initial loading dose of 400 mg followed by a maintenance dose of 200 mg once daily (QD) was selected as the itraconazole dosing regimen in this study.
  Based on the predicted proportion of plasma exposure of metabolites from previous mass balance studies and combined with the previously established safety profile of Rocbrutinib, potent CYP3A inhibition is expected to potentially significantly increase the plasma concentration of Rocbrutinib when co-administered. Therefore, the clinically confirmed minimum effective dose of Rocbrutinib (100 mg) was chosen for co-administration
  Interventions: Drug: Rocbrutinib tablets; Drug: Itraconazole capsules
- Inducer Group (Experimental): The Inducer Group was designed to investigate the drug-drug interaction between Rocbrutinib and rifampicin (a potent CYP3A inducer and P-gp inhibitor). Rifampicin is a recommended potent index CYP3A inducer for clinical studies in the ICH-M12 Guideline on Drug Interactions. The maximum dose and shortest dosing interval in its clinically recommended regimen is 600 mg once daily (QD), so 600 mg QD was selected as the rifampicin dosing regimen in this study.
  Potent CYP3A inducers are expected to either decrease the plasma concentration of Rocbrutinib or have no significant effect on it. Therefore, the clinically recommended higher dose of Rocbrutinib (200 mg) was chosen for co-administration with rifampicin in the Inducer Group.
  In Cycle 2, Rocbrutinib administration was initiated on Day 10 (the 7th day after the start of continuous rifampicin dosing) and continued until the day before the last blood collection for Rocbrutinib (Day 12), which was sufficient to cover the in vivo drug meta
  Interventions: Drug: Rocbrutinib tablets; Drug: Rifampicin capsules

INTERVENTIONS:
Drug: Rocbrutinib tablets — Dosage form: tablets Specification: 100 mg Dosage and administration: 100mg or 200mg, single dose, taken on the designated day according to the treatment plan.
  Dosage schedule: Depending on the cohort, subjects will need to take Rocbrutinib 2 times (inhibitor cohort) or 3 times (inducer cohort) during the study period.
Drug: Itraconazole capsules — Dosage form: Capsules Specifications: 0.1g Dosage and administration: Take 400 mg (4*100 mg capsules) on Day 5, followed by 200 mg (2 100 mg capsules) once daily (QD) from Day 6 to Day 12.
  Duration of medication: The medication was administered for a total of 8 days during the study period.
  Arms: Inhibitor Group
Drug: Rifampicin capsules — Dosage form: Capsules Specifications: 0.15g Dosage and administration: Day 4-Day 12, take 600 mg (4 150 mg capsules) once daily (QD).
  Duration of medication: The medication was administered for a total of 9 days during the study period.
  Arms: Inducer Group

SUMMARY:
This is a phase I, open-label, two-part, fixed-sequence drug interaction study conducted to evaluate the effects of concomitant use of the potent CYP3A4 inhibitor itraconazole or the CYP3A4 inducer rifampin on the pharmacokinetics of Rocbrutinib in healthy subjects.

DETAILED DESCRIPTION:
This study evaluated the changes in the pharmacokinetic profiles of Rocbrutinib under maximal CYP3A inhibition and induction conditions by investigating the co-administration of Rocbrutinib with potent CYP3A inhibitors or inducers at steady state, compared with Rocbrutinib administered alone.

To assess the potential clinical inhibition of OATP1B by Rocbrutinib, blank plasma samples were collected prior to Rocbrutinib administration and 24-hour plasma samples were collected post-administration. The concentration of coproporphyrin I (CP-I) in these samples was detected and analyzed.

Furthermore, the effect of P-gp inhibitors on the drug absorption of Rocbrutinib (when acting as a substrate) was evaluated by investigating two scenarios: co-administration of a single dose of Rocbrutinib with a single dose of the P-gp inhibitor rifampicin, and co-administration of a single dose of Rocbrutinib with the P-gp inhibitor itraconazole at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had no history of serious digestive system (such as inflammatory bowel disease, chronic diarrhea, Crohn's disease, autonomic dysfunction affecting gastric emptying), nervous system, cardiovascular system, genitourinary system, respiratory system, metabolic and endocrine system, musculoskeletal system, hematologic system diseases, or tumors
* Subjects must agree to complete abstinence or use effective physical contraception (including sterilization, intrauterine device or barrier contraception) from the time of signing the informed consent form until 90 days after the last dose of medication, and have no plans to donate sperm or eggs during this period; if female subjects are using hormonal contraceptives, they must stop using them >14 days before the first dose and use at least one of the above contraceptive methods.
* Must be between 18 and 45 years old (inclusive) and be male or female when signing the informed consent form.
* Males weighing ≥50.0 kg or females weighing ≥45.0 kg, with a Body Mass Index (BMI) between 18.0 and 28.0 kg/m² (inclusive). BMI = weight (kg) / height² (m²).
* Able to understand and comply with the requirements of the research plan.
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Abnormalities in screening tests, such as vital signs, physical examination, or laboratory tests are clinically significant and may increase the risk of participants participating in the study or affect the scientific validity of the study.
* Abnormal electrocardiogram or myocardial enzyme levels that are clinically significant as determined by a clinician include, but are not limited to: QTcF ≥ 450 ms (corrected using the Fridricia formula, QTcF = QT/RR1/3, RR = 60/HR), etc.
* The test results for at least one of the following are positive: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, and syphilis-specific antibody.
* Patients who have taken the investigational drug within 4 weeks prior to or are required to take any drugs known to alter liver enzyme activity during the study period.
* The patient must have used any systemic medications (including any vaccines, prescription drugs, over-the-counter drugs, and traditional Chinese medicines), special medical purpose foods, or health supplements within two weeks prior to taking the investigational drug.
* Had consumed foods known to alter liver enzyme activity (such as grapefruit, star fruit, dragon fruit, and their fruit juices) and tobacco (including e-cigarettes) within one week prior to taking the investigational drug.
* Consume any food or beverage containing caffeine, tea, alcohol, or xanthine within 24 hours prior to taking the investigational drug.
* Difficulty swallowing or any condition that affects drug absorption, distribution, metabolism, or excretion.
* Women with childbearing potential who have a positive pregnancy test result or who are currently breastfeeding.
* Those with a history of smoking (smoking more than 5 cigarettes/day within 3 months prior to screening) or who tested positive for nicotine screening.
* Those with a history of alcohol abuse (consuming more than 14 drinks per week, each drink equivalent to 360 ml of beer, 150 ml of wine, or 50 ml of spirits), or those who test positive for alcohol in a breathalyzer test.
* Those with a history of drug abuse/use, or who test positive in drug abuse screening.
* Those with a known history of any allergic reaction requiring medication (including allergic reactions to drugs or food) or who have an allergic disease.
* Individuals who have donated blood or lost ≥400 ml of blood within the three months prior to screening, or those who plan to donate blood during the study period and within three months after its completion, will be considered.
* Those who have undergone surgery within the past 6 months or are expected to require surgery or hospitalization during the study period will be screened.
* Candidates who have participated in other drug or medical device clinical trials within the three months prior to screening, or who plan to participate in other drug or medical device clinical trials during the study period, are eligible to be screened.
* Subjects with special dietary requirements or who are expected to be unable to comply with the research center's dietary requirements during their hospitalization
* The researchers believe that there are other circumstances that make the participants unsuitable to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
AUC | Until 72 hours or 96 hours after Rocbrutinib
  Area under the curve
Cmax | Until 72 hours or 96 hours after Rocbrutinib
  Plasma peak concentration of Rocbrutinib
t1/2 | Until 72 hours or 96 hours after Rocbrutinib
  Terminal phase half-life of Rocbrutinib

SECONDARY OUTCOMES:
Plasma coprophyrin I (CP-I) concentration | Baseline and 24 hours after Rocbrutinib
  Plasma coprophyrin I (CP-I) concentration
Adverse events | Up to 20 days after Rocbrutinib
  Adverse events were evaluated by investigators based on clinical examination findings and observations in accordance with the CTCAE Version 5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Since this is a clinical pharmacology study enrolling healthy subjects, it is planned to report the study results through peer-reviewed publications, and individual participant data will not be shared.